CLINICAL TRIAL: NCT05188716
Title: Investigating Mechanisms That Dictates Tumor Immunogenicity and Exploring Biomarkers That Could Help Predict the Anti-tumor Immune Response in Patients With Cervical Cancer
Brief Title: Mechanisms and Biomarkers for Tumor Immunogenicity Modulation in Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Chuangzhen Chen (Other)
Responsible Party: Sponsor-Investigator, Chuangzhen Chen, Deputy Director, Department of Radiation Oncology, Shantou University Medical College
Organization: Shantou University Medical College (Other)
Other Study IDs: Immune002
Record Dates: First submitted 2021-05-20; First posted 2022-01-12 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer; Benign Tumor of Uterus
Keywords: Cervical cancer; Tumor immunogenicity
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples or the epithelium of cervix or other biological samples will be obtained from patients receiving surgery. For patients who will be treated with definite chemoradiotherapy, tumor samples, blood samples and microbiota will be collected before and during the course of treatment, and when the disease progressed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate mechanisms that dictate tumor immunogenicity and to explore potential biomarkers that could help predict changes of tumor immunogenicity and therapeutic response in patients with cervical cancer after chemoradiotherapy or surgery.

DETAILED DESCRIPTION:
Patients pathologically confirmed with cervical cancer or benign gynecologic tumor that requires chemoradiotherapy or surgery will be recruited to this study. Tumor samples, normal epithelium of the cervix or other biological samples will be obtained from patients who will receive surgery to establish the baseline status of tumor/mucosal immunogeneicity. For patients undergoing definite radiotherapy, tumor biopsies, collection of blood samples and microbiota will be performed before and during the course of treatment and when the disease progressed. These biological specimens will be used to investigate signaling pathways that determine tumor immungenenicity and their dynamic changes during treatment and to explore feasible biomarkers that could reflect and help monitor the inter- and intra-patient varariation of tumor immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Pathological proven diagnosis of cervical cancer or benign gynecologic tumor and will undergoing panhysterectomy or pathological proven diagnosis of cervical cancer and will undergoing radiotherapy
* Tumor accessible for biopsy during the course of radiotherapy or tumor samples could be obtained via surgery
* Patient must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* History of autoimmune diseases
* History of immunotherapy
* History of pelvic radiotherapy
* Will receive immunotherapy during the course of treatment
* Contraindications for biopsy, such as high bleeding risk

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients proven diagnosis of cervical cancer or benign gynecologic tumor and will have radiotherapy as part of their therapeutic regimens or will undergo surgery in Cancer Hospital of Shantou University Medical College.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Expression status of biomarkers during treatment and follow-up | From the date of enrollment until the date of disease progression, assessed up to 5 years
  Expression status of biomarkers in patients' biological specimens through the course of treatment and during follow-up as assessed by a variety of means, including RNA-seq, DNA-seq, RT-qPCR, IHC, WB, flow cytometry and ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Chuangzhen Chen, MD, Principal Investigator — Affiliated Cancer Hospital of Shantou University Medical College
Locations (1):
- Cancer Hospital of Shantou University Medical College, Shantou, Guangdong, China